CLINICAL TRIAL: NCT06239909
Title: Clinical Outcomes of the Adjustable Artificial Sphincter Victo in the Treatment of Male Incontinence Due to Prostate Surgery - Prospective Follow-up Study
Brief Title: Adjustable Artificial Sphincter Victo in the Treatment of Male Incontinence Due to Prostate Surgery
Status: Recruiting | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: AUS-V-001
Record Dates: First submitted 2024-01-12; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence; artificial urinary sphincter; pad-weight test; quality of life
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Urinary incontinence due to prostate surgery: Consecutive adult male patients with urinary incontinence due to prostate surgery.
  Interventions: Other: 24-h pad-weight test; Other: Patient Global Impression - Improvement Questionnaire

INTERVENTIONS:
Other: 24-h pad-weight test — The patients will be asked to perform the 24-h pad-weight test
Other: Patient Global Impression - Improvement Questionnaire — The patient-reported outcome, as measured by PGI-I (Patient Global Impression - Improvement Questionnaire)

SUMMARY:
The aim of this prospective academic research study is to evaluate the efficacy and safety of the Victo adjustable artificial sphincter in the treatment of male patients with urinary incontinence due to prostate surgery.

DETAILED DESCRIPTION:
This is a non-interventional prospective study. The study will include male patients who underwent the Victo artificial sphincter placement due to severe incontinence.

Before the procedure, all patients will undergo a standard diagnostic work-up. After the procedure, the patients will be invited for regular visits 3 months after device activation and subsequently every 12 months. In addition to the regular visits, patients will be allowed to contact the study center at any time if their continence worsens enough to require adjustment or if they experience any complications.

The surgical technique of the Victo artificial sphincter implantation has been described in detail elsewhere.

A non-parametric one-way ANOVA Friedman test will be used to compare the changes of categorical variables from baseline to the end of follow-up. Wilcoxon rank-sum test will be used to assess the change of the non-categorical variables. P-value < 0.05 is considered statistically significant and no correction for multiple testing will be applied.

ELIGIBILITY:
Inclusion Criteria:

* urinary incontinence due to previous prostate surgery
* primo-implantation of the artificial urinary sphincter
* subject willing and able to give informed consent

Exclusion Criteria:

- none

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Study Population: Patients with moderate to severe incontinence due to previous prostate surgery, seeking medical help (implantation of the artificial urinary sphincter)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Severity of incontinence as measured using 24-hour pad-weight test (24PWT) | 72 hours
  The severity of incontinence will be measured using the 24PWT. The patients will be asked to perform the test three times, and the average weight of the three measurements will be recorded. The change in severity of incontinence as measured by 24PWT will be observed from baseline to the end of observation.

SECONDARY OUTCOMES:
Patients-reported outcomes of treatment | 5 years
  The patients-reported outcomes will be measured using the Patient Global Impression of Improvement (PGI-I) index. The Patient Global Impression of Improvement (PGI-I) is a global index that may be used to rate the response of a condition to a therapy. The PGI-I is a transition scale that is a single question asking the patient to rate their urinary tract condition now, as compared with how it was prior to beginning treatment on a scale from 1. (Very much better) to 7. (Very much worse).
Treatment safety assessment | 5 years
  The safety of treatment will be measured by evaluation of the reported treatment-related complications using the Clavien-Dindo classification. The Clavien-Dindo system is widely used throughout surgery for grading adverse events (i.e. complications) which occur as a result of surgical procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Krhut, prof.,MD, PhD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

REFERENCES:
- [Background] Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont). 2007 Jul;4(7):28-37. PMID 20526405
- [Background] Weibl P, Hoelzel R, Rutkowski M, Huebner W. VICTO and VICTO-plus - novel alternative for the mangement of postprostatectomy incontinence. Early perioperative and postoperative experience. Cent European J Urol. 2018;71(2):248-249. doi: 10.5173/ceju.2018.1655. Epub 2018 Apr 19. No abstract available. PMID 30038818
- [Background] Krhut J, Zachoval R, Smith PP, Rosier PF, Valansky L, Martan A, Zvara P. Pad weight testing in the evaluation of urinary incontinence. Neurourol Urodyn. 2014 Jun;33(5):507-10. doi: 10.1002/nau.22436. Epub 2013 Jun 24. PMID 23797972